CLINICAL TRIAL: NCT04329949
Title: A Phase 3 Study of Relacorilant in Combination With Nab-Paclitaxel in Patients With Metastatic Pancreatic Ductal Adenocarcinoma (RELIANT)
Brief Title: Study of Relacorilant in Combination With Nab-Paclitaxel in Patients With Metastatic Pancreatic Ductal Adenocarcinoma
Acronym: RELIANT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The independent data monitoring committee found no safety issues, however the observed response rate did not meet the predefined threshold for continuing the study. The study was terminated by the Sponsor.
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CORT125134-553
Record Dates: First submitted 2020-03-13; First posted 2020-04-01 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Cancer; mPDAC; Metastatic Pancreatic Ductal Adenocarcinoma; Glucocorticoid Receptor; Nab-paclitaxel; GR Antagonist; Relacorilant; Abraxane
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — relacorilant; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Relacorilant with nab-paclitaxel (Experimental): Patients will be treated with relacorilant, administered orally, once daily in combination with nab-paclitaxel on Days 1, 8, and 15 of each 28-day cycle.
  Interventions: Drug: Relacorilant, 100 mg and 25 mg; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Relacorilant, 100 mg and 25 mg — Relacorilant is supplied as capsules for oral dosing.
  Other Names: CORT125134
Drug: Nab-paclitaxel — Nab-paclitaxel is administered as IV infusion over 30 minutes on Days 1, 8, and 15 of each 28-day cycle.
  Other Names: Abraxane

SUMMARY:
This is a Phase 3, open-label study to evaluate the objective response rate (ORR), in patients with metastatic pancreatic ductal adenocarcinoma (mPDAC) treated with relacorilant in combination with nab-paclitaxel, according to blinded independent central review.

DETAILED DESCRIPTION:
Relacorilant is a small-molecule antagonist of the glucocorticoid receptor (GR). The goals of this study are to evaluate the efficacy, safety, and pharmacokinetics (PK) of relacorilant in combination with nab-paclitaxel in the treatment of metastatic pancreatic ductal adenocarcinoma.

Eligible patients are those with mPDAC who have received at least 2 prior lines of therapy for pancreatic ductal adenocarcinoma in any setting, including at least 1 prior gemcitabine-based therapy and at least 1 prior fluoropyrimidine-based therapy.

Patients will receive treatment until progressive disease (PD) (per RECIST v1.1) as determined by the Investigator, experiencing unmanageable toxicity, or until other treatment discontinuation criteria are met. All patients will be followed for documentation of disease progression and survival information (i.e., date and cause of death) and subsequent treatment.

ELIGIBILITY:
Inclusion Criteria - Patients must have the following:

Histologically confirmed PDAC with metastatic disease

Received at least 2 prior lines of therapy for PDAC in any setting, including at least 1 prior gemcitabine-based therapy and at least 1 prior fluoropyrimidine-based therapy

Received no more than 4 prior lines of cytotoxic or myelosuppressive therapy for PDAC

A measurable lesion at baseline (within 21 days prior to the first dose of relacorilant) per RECIST v1.1, as assessed by the Investigator

Willingness to provide blood samples and tumor tissue (primary or metastatic) for research purposes

Karnofsky performance status (KPS) score of ≥70

Adequate gastrointestinal absorption. If the patient has undergone gastric bypass surgery and/or surgery of gastrointestinal or hepatobiliary tract, the patient must demonstrate adequate absorption as evidenced by albumin ≥3.0 g/dL, controlled pancreatic insufficiency (if present), and lack of evidence of malabsorption

Adequate organ and marrow function (determined through blood and urine tests)

Exclusion Criteria - Patients must not have the following:

Pancreatic neuroendocrine tumors, lymphoma of the pancreas, acinar pancreatic cancer, or ampullary cancer

Known untreated parenchymal brain metastasis or have uncontrolled central nervous system metastases. Patients must not require steroids and must be neurologically stable without corticosteroids for a minimum of 3 weeks prior to Cycle 1 Day 1

Clinically relevant toxicity from prior systemic cytotoxic therapies or radiotherapy that in the opinion of the Investigator has not resolved to Grade 1 or less prior to enrollment, including peripheral neuropathy that is ongoing and greater than Grade 1 in severity, according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0

History of hypersensitivity or severe reaction to either relacorilant or nab-paclitaxel, or to similar classes of either drug

Taken the following medications prior to enrollment:

1. An investigational product, cytotoxic chemotherapy, or targeted agent within 14 days
2. Radiotherapy within 21 days
3. Palliative radiotherapy within 1 week of Cycle 1 Day 1, or if toxicities from radiotherapy are Grade 2 severity or higher or have not recovered to baseline
4. Systemic or prescription-strength topical corticosteroids for the purposes of treating a chronic nononcologic indication within 21 days.

Requirement for treatment with chronic or frequently used oral or inhaled corticosteroids for medical conditions or illnesses (e.g., rheumatoid arthritis, asthma, or immunosuppression after organ transplantation)

Taking a concomitant medication that is a strong CYP3A (cytochrome P450 3A) or CYP2C8 inhibitor or inducer, or a substrate of CYP3A or CYP2C8 and has a narrow therapeutic window

Concurrent treatment with mifepristone or other GR antagonists

Any clinically significant uncontrolled condition(s) or any medical condition which in the opinion of the Investigator places the patient at an unacceptably high risk for toxicities or impair study participation or cooperation

Any major surgery within 21 days prior to enrollment

Endoscopic retrograde cholangiopancreatography with persistence of any of the following:

1. Bilirubin ≥1.5 × ULN (Upper Limit of Normal)
2. Amylase >2 × ULN and abdominal pain or amylase >3 × ULN (with or without symptoms)
3. Fever or signs of infection
4. Decreasing hemoglobin or signs of blood loss.

A history of human immunodeficiency virus (HIV) or current chronic/active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV). (Patients with chronic or active hepatitis B as diagnosed by serologic tests are excluded from the study. In equivocal cases, hepatitis B or C polymerase chain reaction results may be performed and must be negative for enrollment.)

A rapid decline in KPS score or serum albumin (≥20%), or have progressive pain symptoms indicative of rapid clinical deterioration, in the opinion of the Investigator, prior to enrollment. These patients will become ineligible if rapid decline is observed during the screening period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Guyer, PharmD, Study Director — Corcept Therapeutics, Menlo Park, CA 94025
Locations (18):
- United States (18):
  - Site #038, Scottsdale, Arizona
  - Site #171, Duarte, California
  - Site #076, Los Angeles, California
  - Site #032, Aurora, Colorado
  - Site #009, Atlanta, Georgia
  - Site #184, Goshen, Indiana
  - Site #065, Baltimore, Maryland
  - Site #058, Detroit, Michigan
  - Site #185, Omaha, Nebraska
  - Site #182, Buffalo, New York
  - Site #044, New York, New York
  - Site #222, New York, New York
  - Site #077, Columbus, Ohio
  - Site #186, Toledo, Ohio
  - Site #172, Pittsburgh, Pennsylvania
  - Site #175, Knoxville, Tennessee
  - Site #176, Nashville, Tennessee
  - Site #173, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 18 study sites in the United States.
Groups:
- Relacorilant With Nab-paclitaxel: Patients were treated with relacorilant, administered orally, once daily in combination with nab-paclitaxel on Days 1, 8, and 15 of each 28-day cycle.
  Relacorilant, 100 mg and 25 mg: Relacorilant was supplied as capsules for oral dosing.
  Nab-paclitaxel: Nab-paclitaxel was administered as IV infusion over 30 minutes on Days 1, 8, and 15 of each 28-day cycle.
Period: Overall Study
Arm/Group | Relacorilant With Nab-paclitaxel
Started | 43
Completed | 0
Not Completed | 43
Not completed — Death | 36
Not completed — Withdrawal by Subject | 4
Not completed — Termination of study by sponsor | 3

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Arm/Group | Relacorilant With Nab-paclitaxel
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.2 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 35
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Blinded Independent Central Review (BICR)
Description: Percentage of patients with measurable disease at baseline who achieved confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, as assessed by Blinded Independent Central Review (BICR). Tumor assessment consisted of computerized tomography (CT) scan or, with Sponsor approval, magnetic resonance imaging (MRI). CR was defined as disappearance of all target lesions; any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm. PR was defined as ≥30% decrease in the sum of the diameters (SOD) of target lesions.
Time Frame: Baseline and up to 32 weeks
Population: Intent-to-Treat (ITT) Population: Patients enrolled and treated with at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant With Nab-paclitaxel
Number analyzed (Participants) | 43
Participants
  Complete response | 0
  Partial response | 0
  No response | 43

2. Secondary Outcome: Objective Response Rate (ORR) Per Investigator Assessment
Description: Percentage of patients with measurable disease at baseline who achieved confirmed CR or PR per RECIST v1.1, as assessed by the Investigator. Tumor assessment consisted of CT scan or, with Sponsor approval, MRI. CR was defined as disappearance of all target lesions; any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm. PR was defined as ≥30% decrease in the SOD of target lesions.
Time Frame: Baseline and up to 48 weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant With Nab-paclitaxel
Number analyzed (Participants) | 43
Participants
  Complete response | 0
  Partial response | 0
  No response | 43

3. Secondary Outcome: Best Overall Response (BOR)
Description: To evaluate the best overall response of CR, PR, stable disease (SD), or PD per RECIST v1.1. as assessed by BICR. Tumor assessment consisted of CT scan or, with Sponsor approval, MRI. CR was defined as disappearance of all target lesions; any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm. PR was defined as ≥30% decrease in the SOD of target lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD was defined as ≥20% increase in the SOD of target lesions or the appearance of one or more new lesions.
Time Frame: Baseline and up to 32 weeks
Population: Evaluable Population: Patients in the ITT population who had at least 1 post-baseline radiographic tumor assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant With Nab-paclitaxel
Number analyzed (Participants) | 31
Participants
  Complete response | 0
  Partial response | 0
  Stable disease | 20
  Progressive disease | 10
  Non-evaluable | 1

4. Secondary Outcome: Duration of Response (DOR)
Description: To evaluate the duration of response as the time of objective response (CR or PR) to the time of disease progression or death, per RECIST v1.1 as assessed by BICR and the Investigator. Tumor assessment consisted of CT scan or, with Sponsor approval, MRI. CR was defined as disappearance of all target lesions; any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm. PR was defined as ≥30% decrease in the SOD of target lesions. PD was defined as ≥20% increase in the SOD of target lesions or the appearance of one or more new lesions.
Time Frame: Time of response up to 32 weeks
Population: This outcome was not analyzed because the response rate was 0%.
Arm/Group | Relacorilant With Nab-paclitaxel
Number analyzed (Participants) | 0

5. Secondary Outcome: Disease Control Rate (DCR)
Description: To evaluate patients disease control rate of CR, PR, or SD at 18 weeks, per RECIST v1.1 as assessed by the Investigator. Tumor assessment consisted of CT scan or, with Sponsor approval, MRI. CR was defined as disappearance of all target lesions; any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm. PR was defined as ≥30% decrease in the SOD of target lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Enrollment through 18 weeks
Population: Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant With Nab-paclitaxel
Number analyzed (Participants) | 31
Participants | 5

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: To evaluate PFS as median time to disease progression per RECIST v1.1, or death, as assessed by BICR. Tumor assessment consisted of CT scan or, with Sponsor approval, MRI. Disease progression was defined as ≥20% increase in the SOD of target lesions or the appearance of one or more new lesions.
Time Frame: Baseline and up to 31 weeks.
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Relacorilant With Nab-paclitaxel
Number analyzed (Participants) | 43
Months | 2.4 [1.4 to 4.2]

7. Secondary Outcome: Overall Survival (OS)
Description: To evaluate OS as median time to death by any cause.
Time Frame: Baseline and up to 70 weeks
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Relacorilant With Nab-paclitaxel
Number analyzed (Participants) | 43
Months | 3.9 [2.8 to 4.9]

8. Secondary Outcome: Progression-Free Survival (PFS)
Description: To evaluate PFS as the percentage of patients who are progression-free at 3, 6, and 12 months per RECIST v1.1, as assessed by BICR. Tumor assessment consisted of CT scan or, with Sponsor approval, MRI. Disease progression was defined as ≥20% increase in the SOD of target lesions or the appearance of one or more new lesions.
Time Frame: Enrollment through 3 months, 6 months, and 12 months
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relacorilant With Nab-paclitaxel
Number analyzed (Participants) | 43
Percentage of participants
  3 months | 44.77 [28.97 to 59.38]
  6 months | 8.00 [1.57 to 21.50]
  12 months | NA [NA to NA] — The Kaplan-Meier estimates and corresponding 95% confidence interval (CI) for the Progression-Free Survival (PFS) Rates at Months 3, 6, and 12 are provided. Due to no subjects being progression-free by Month 12, the PFS rate and 95% CI at that timepoint are not estimable and shown as NA.

9. Secondary Outcome: Overall Survival (OS)
Description: To evaluate OS as the percentage of patients surviving at 3, 6, and 12, months.
Time Frame: Enrollment through 3 months, 6 months, and 12 months
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relacorilant With Nab-paclitaxel
Number analyzed (Participants) | 43
Percentage of participants
  3 months | 64.12 [47.65 to 76.61]
  6 months | 21.55 [10.23 to 35.58]
  12 months | 10.77 [3.44 to 22.91]

10. Secondary Outcome: Cancer Antigen (CA)19-9
Description: To assess cancer antigen 19-9 (CA19-9) response at 8 and 16 weeks in patients who have elevated CA19-9 at baseline. Response was defined as ≥50% reduction in CA19-9.
Time Frame: Enrollment through 8 weeks and 16 weeks
Population: Patients in the ITT population who had elevated CA19-9 at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant With Nab-paclitaxel
Number analyzed (Participants) | 39
Participants
  8 weeks | 5
  16 weeks | 3

11. Secondary Outcome: Tumor Response Per European Organization for Research and Treatment of Cancer (EORTC) Criteria
Description: To assess tumor response based on changes in fluorodeoxyglucose-positron emission tomography (FDG-PET) scan at 6 weeks per the EORTC criteria, as assessed by BICR.
Time Frame: Enrollment through 6 weeks
Population: Patients in the ITT Population with measurable disease at baseline by FDG-PET evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant With Nab-paclitaxel
Number analyzed (Participants) | 23
Participants
  Complete metabolic response | 0
  Partial metabolic response | 6
  Stable metabolic disease | 9
  Progressive metabolic disease | 8

12. Secondary Outcome: Time to Progression (TTP)
Description: To evaluate TTP as median time to disease progression per RECIST v1.1, as assessed by the Investigator. Tumor assessment consisted of CT scan or, with Sponsor approval, MRI. Disease progression was defined as ≥20% increase in the SOD of target lesions or the appearance of one or more new lesions.
Time Frame: Baseline and up to 32 weeks
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Relacorilant With Nab-paclitaxel
Number analyzed (Participants) | 43
Months | 4.2 [1.6 to NA] — The upper 95% confidence interval of median TTP was not calculable due to insufficient number of patients with events.

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study treatment (up to 73 weeks)
Arm/Group | Relacorilant With Nab-paclitaxel
All-Cause Mortality (participants affected / at risk) | 36/43
Serious Adverse Events (participants affected / at risk) | 23/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relacorilant With Nab-paclitaxel (N=43)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 2
Obstruction gastric (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Pyrexia (General disorders) | 1
Sepsis (Infections and infestations) | 3
Bacteraemia (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Device occlusion (Product Issues) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Relacorilant With Nab-paclitaxel (N=43)
Anaemia (Blood and lymphatic system disorders) | 13
Neutropenia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 3
Tachycardia (Cardiac disorders) | 3
Nausea (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 14
Abdominal pain (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 9
Ascites (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 6
Dry mouth (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 34
Oedema peripheral (General disorders) | 9
Mucosal inflammation (General disorders) | 4
Fall (Injury, poisoning and procedural complications) | 3
Neutrophil count decreased (Investigations) | 12
White blood cell count decreased (Investigations) | 9
Platelet count decreased (Investigations) | 8
Weight decreased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 17
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12
Hypokalaemia (Metabolism and nutrition disorders) | 10
Hyponatraemia (Metabolism and nutrition disorders) | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 3
Confusional state (Psychiatric disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 5
Hypotension (Vascular disorders) | 6

LIMITATIONS AND CAVEATS:
The independent data monitoring committee found no safety issues, however the observed response rate did not meet the predefined threshold for continuing the study. The study was terminated by the Sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual publications will be allowed before publication of the multicenter results except as agreed with the Sponsor. The Investigator agrees to submit all manuscripts or abstracts to the Sponsor for review before submission to the publisher. The Sponsor will comply with the requirements for publication of study results and determination of authorship in accordance with standard editorial and ethical practice and with the International Committee of Medical Journal Editors requirements.

DOCUMENTS (2):
  • Study Protocol (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT04329949/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT04329949/SAP_001.pdf